CLINICAL TRIAL: NCT02360865
Title: Mechanisms of Exercise Intolerance in Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-2-2013-150 - project 2
Record Dates: First submitted 2015-01-19; First posted 2015-02-11 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD (Experimental): Acute exercise bouts
  Interventions: Other: Exercise
- Healthy (Active Comparator): Acute exercise bouts
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
1: Is endothelium function impaired in COPD? Other chronic cardiovascular diseases are associated with endothelial dysfunction, and the endothelium plays an important role in regulating vascular tone, tissue blood flow, coagulation and the inflammation process. Although the specific causes of endothelial dysfunction remain unclear, physical inactivity, chronic systemic inflammation and smoking are all known to be associated with endothelial abnormality.

2. Is Muscular Sympathetic Nerve Activity (MSNA) increased in COPD? A balanced regulation of blood flow to skeletal muscles may be disturbed by pathophysiology and may therefore contribute to the exercise intolerance and skeletal muscle depletion seen in patients with COPD.Skeletal muscle blood flow is tightly regulated to match tissue oxygen demands and is thus adapted to meet energy requirements. During physical activity, the sympathetic nervous system is activated ("exercise pressor reflex"), resulting in increased ventilation, heart rate and a redistribution of cardiac output from inactive to active tissues. The redistribution of cardiac output to the body organs is heterogeneous. Blood flow to skeletal, respiratory and cardiac muscle increases as exercise intensity increases, whereas blood flow to gastrointestinal, renal and reproductive tissues decreases. As blood pressure during exercise remains largely unchanged, the redistribution of blood flow is caused by changes in vascular conductance. These conductance changes are caused by an overall vasoconstriction induced by the increased sympathetic outflow of noradrenaline (NA), and a vasodilation of vascular beds supplying the working skeletal -, cardiac- and respiratory muscle.

ELIGIBILITY:
Inclusion Criteria:

* Forced Expiratory Volume at on second/ Forced Vital Capacity fixed ratio <0.70, - Forced Expiratory Volume at one second <60% of predicted and Medical
* Research Council scale > or equal to 3
* Arterial oxygen saturation at rest> 90%,
* Body Mass Index >18,
* Left Ventricle Ejection Fraction> 45.

Exclusion Criteria:

* Unstable ischemic heart disease,
* severe heart valve failure,
* pulmonary emboli,
* severe heart failure,
* severe infections,
* musculoskeletal disorders,
* malignant disease,
* contraindicated medicine as anticoagulants.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Endothelium function during acute exercise (one legged kicking) by Flow doppler | On one experimental day during acute exercise (one legged knicking) and change from baseline
  Flow doppler
Muscular Sympathetic Nerve Activity During acute exercise (handgrip and leg isometric leg extension) by Peroneal microneurography | On one experimental day during acute exercise (handgrib and leg isometric leg extension) and change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Physical Activity Research, Copenhagen, Capital Region, Denmark